CLINICAL TRIAL: NCT06537570
Title: The Effect of Guided Imagery Practice on Psychosocial Health and Fear of Childbirth in Primiparous Pregnant Women: A Randomized Controlled Trial
Brief Title: The Effect of Guided Imagery Practice on Psychosocial Health and Fear of Childbirth in Primiparous Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ece Kaplan, Asst. Prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAUN-EBE-EKD-01
Record Dates: First submitted 2024-01-15; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related
Keywords: Fear of childbirth; guided imagery; primiparous pregnant women; psychosocial health
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery Practice (Experimental): Pregnant women in the experimental group were administered pre-tests (Personal Information Form, Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version) just before watching the guided imagery video. In the first interview with pregnant women, video viewing days and hours were determined by giving information about the guided imagery video. Pregnant women were then shown the guided imagery video consisting of a total of 12 weeks, once a day for 15 minutes and 50 seconds. Immediately after the 12-week period was completed, post-tests (Psychosocial Health Evaluation Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version) were administered to the pregnant women.
  Interventions: Behavioral: Guided Imagery Practice
- group (No Intervention): Pregnant women in the control group were administered pre-tests (Personal Information Form, Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale) and post-tests (Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version) 12 weeks later and no practice was performed except routine practices during outpatient follow-up.

INTERVENTIONS:
Behavioral: Guided Imagery Practice — Before the guided imagery application, the language translation of the guided imagery usage steps guide prepared by Owen (2010)27 was done by a translation center in a certified manner. Then, a relaxing, soothing, soft and slow-paced CD consisting of mixed nature sounds, photographs and music lasting 15 minutes and 50 seconds was prepared in the sound recording studio with the psychological counselor.
  Data collection forms were filled in by the researcher using face-to-face interview technique for the women who agreed to participate in the study. The guided imagery video was shared with the women and they were made to watch it once a day for 12 weeks in a quiet, calm, uncrowded, dimly lit room in their homes. The women in the control group did not receive any interventions other than routine interventions during outpatient follow-up.
  Other Names: Guided Imagery
  Arms: Guided Imagery Practice

SUMMARY:
Physical changes that occur during pregnancy, transition to parenthood and taking on new responsibilities cause burden, anxiety and stress in women and negatively affect psychosocial health. One of the conditions that negatively affect psychosocial health during pregnancy is the fear of childbirth. One of the current methods used in the management of the pregnancy process is guided imagery.It is known that guided imagery practice reduces stress and anxiety in pregnant women, increases well-being and is beneficial to their daily lives, contributes positively to mother-baby attachment, and reduces pain in childbirth.

DETAILED DESCRIPTION:
2.1.Study Design

This research was conducted as a randomized controlled experimental study to determine the effect of guided imagery on the psychosocial health and fear of childbirth of primiparous pregnant women. The study was conducted between July 20, 2022 and January 20, 2023 with pregnant women admitted to the obstetrics and gynecology outpatient clinic of XXX Hospital in Gaziantep, Turkey. The hospital where the study was conducted has 7 gynecology outpatient clinics and 1 pregnancy school.

2.2.Sample

The population of the research consisted of all primiparous pregnant women in the 24-28th week of pregnancy. The sample size was calculated using the G Power program. Previous studies were examined and the expected confidence intervals of the "Psychosocial Health Assessment Scale in Pregnancy (PPHAS)" were determined and the confidence interval was calculated as 80 primiparous with α = 0.05, test power (1-β) 0.95, and effect size d= 1.14. Minimum number of pregnant women required in the two groups was found to be 40 for the expectation that there would be a significant difference between the experimental group and the control group in terms of psychosocial health. The sample of the study consisted of 80 pregnant women, 40 in the experimental group and 40 in the control group. The study reached 91 participants, but 11 participants were excluded because they refused to participate in the study (Figure 1). Medcalc version 18.11.3 was used for the randomization list in assigning pregnant women to groups.

Study inclusion criteria of volunteers

1. Volunteer to participate in the study
2. Having no condition to prevent communication
3. Age 18-35
4. No vision and hearing problems
5. At the 24th-28th week of pregnancy
6. With a single fetus
7. Primiparous pregnancies

Study exclusion criteria of volunteers

1. Illiterate
2. Before the 24th week of pregnancy
3. Having multiple pregnancies
4. Multiparous
5. With psychopathological disease
6. Pregnant women with medical or pregnancy complications

2.3.Data Collection

Before the guided imagery application, the language translation of the guided imagery usage steps guide prepared by Owen was done by a translation center in a certified manner. Then, a relaxing, soothing, soft and slow-paced CD consisting of mixed nature sounds, photographs and music lasting 15 minutes and 50 seconds was prepared in the sound recording studio with the psychological counselor.

Data collection forms were filled in by the researcher using face-to-face interview technique for the women who agreed to participate in the study. The guided imagery video was shared with the women and they were made to watch it once a day for 12 weeks in a quiet, calm, uncrowded, dimly lit room in their homes. The women in the control group did not receive any interventions other than routine interventions during outpatient follow-up.

2.4.Data Collection Tools

In this study, data collection tools were prepared by the researcher by reviewing the literature on the subject. Data collection tools consist of three parts (Annex-1):

2.4.1.Personal information form

The content of the personal information form consists of two parts. The first part included questions about the socio-demographic characteristics of pregnant women (age, education level, family type, occupation, and duration of marriage). As for the second part, there were questions about obstetric characteristics (gestational week, information about delivery, miscarriage, and abortion).

2.4.2.Psychosocial Health Assessment Scale in Pregnancy (PPHAS)

The Psychosocial Health Assessment Scale in Pregnancy was developed by Yıldız in 2011 as a scale consisting of six dimensions and 46 items to assess the psychosocial health of pregnant women. In the scale, the first sub-dimension evaluates "Characteristics of pregnancy and spousal relationship", the second sub-dimension evaluates "Characteristics of anxiety and stress", the third sub-dimension evaluates "Characteristics of domestic violence", the fourth sub-dimension evaluates "Characteristics of psychosocial support need", the fifth sub-dimension evaluates "Family characteristics" and the items in the sixth sub-dimension evaluates "Characteristics of physical-psychosocial changes related to pregnancy". In the scale, it is stated that each item should be scored between 1-5 (1= Not at all, 2= A little, 3= Moderately, 4= A lot, 5= Very much). Before calculating the total score, the score calculation of 29 items in the scale should be made by reversing the score calculation and the remaining 17 items should be evaluated as specified. The minimum score that can be obtained from the scale is 46 and the maximum score is 230. The total score obtained from the scale is divided by the number of items to determine the mean value and a result between 1 and 5 is obtained. As a result, as the total score moves away from 5 and approaches 1, it indicates that there is a problem at that level in psychosocial health during pregnancy, and a score of 1 indicates that psychosocial health is very poor. In the validity and reliability study of the scale, Cronbach's alpha reliability coefficient was found to be 0.93.29 In this study, Cronbach's alpha reliability coefficient was found to be 0.84.

The score ranges in the evaluation of the PPHAS are as follows;

* ≤ 1.79 Very low (very bad)
* 1.80 - 2.79 Low (bad)
* 2.80 - 3.39 Medium
* 3.40 - 4.19 Good
* 4.20 ≤ Very good

2.4.3.Wijma Birth Expectation/ Experience Scale-A Version (W-DEQ/ A Version)

It was developed by Wijma et al. (1988) to measure the fear of childbirth experienced by women. The scale consists of 33 items. The answers in the scale are numbered from 0 to 5 and are six-point Likert type. 0 is expressed as "completely" and 5 is expressed as "none". While the minimum score on the scale is 0, the maximum score is 165. As the score increases, the fear of childbirth experienced by women increases. It is calculated by reversing 14 questions. The clinical level of fear is 85 and above. The scale, which was adapted into Turkish by Körükcü et al. (2008) and its validity and reliability was performed, has a Cronbach's alpha value of 0.89 and Split-half reliability of 0.91.30 In this study, Cronbach's alpha reliability coefficient was found to be 0.79.

Score ranges for the evaluation of Version A (W-DEQ) are as follows;

* W-DEQ score ≤37: indicates mild level fear ,
* W-DEQ score = 38-65: indicates moderate level fear,
* W-DEQ score = 66-84: indicates severe level fear,
* W-DEQ score ≥85: indicates clinical level fear.6

2.5.Initiative

After interviewing the women who met the inclusion criteria, the purpose of the study was explained and written informed consent was obtained from those who agreed to participate in the study. The interventions are shown in the flow plan of the study (Figure 2).

2.5.1.Procedures Applied to the Study Group

Pregnant women in the experimental group were administered pre-tests (Personal Information Form, Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version (W-DEQ/ A Version)) just before watching the guided imagery video. In the first interview with pregnant women, video viewing days and hours were determined by giving information about the guided imagery video. Pregnant women were then shown the guided imagery video consisting of a total of 12 weeks, once a day for 15 minutes and 50 seconds. Immediately after the 12-week period was completed, post-tests (Psychosocial Health Evaluation Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version (W-DEQ/ A Version)) were administered to the pregnant women.

2.5.2.Procedures Applied to Control Group

Pregnant women in the control group were administered pre-tests (Personal Information Form, Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version (W-DEQ/ A Version)) and post-tests (Psychosocial Health Assessment Scale in Pregnancy and Wijma Birth Expectancy/ Experience Scale - A Version (W-DEQ/ A Version)) 12 weeks later and no practice was performed except routine practices during outpatient follow-up.

2.6.Analysis

The data obtained from this study were coded by the researcher and then transferred to the SPSS for Windows 26.0 (IBM Corp., Armonk, NY, USA) computer program and the necessary analyses were made in this program. Shaphiro wilk test was applied to determine whether the scores of the pregnant women from the scales showed normal distribution. In the comparison of numerical variables in 2 independent groups, data with normal distribution were analyzed by Student t test. One-factor ANOVA for dependent samples was used to determine the effect of guided imagery on PPHAS and W-DEQ/ A. Effect sizes were calculated with partial Eta squared (ηp2), and if they were calculated between 00 and .30, they were considered very low; if they were between .30 and .50, they were considered low; If they were between .50 and .70, they were considered moderate, if they were between .70 and .90, they were considered high; if they were between .90 and 1.00, they were considered very high.31 Paired Sample t-test was used for the pre-test and post-test comparison of the subscales of PPHAS and W-DEQ/ A in the dependent group. The significance level was taken as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Having no condition to prevent communication
* Age 18-35
* No vision and hearing problems
* At the 24th-28th week of pregnancy
* With a single fetus
* Primiparous pregnancies

Exclusion Criteria:

* Illiterate
* Before the 24th week of pregnancy
* Having multiple pregnancies
* Multiparous
* With psychopathological disease
* Pregnant women with medical or pregnancy complications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Psychosocial Health Assessment Scale in Pregnancy | 12 weeks
  Psychosocial Health Assessment Scale in Pregnancy. The minimum score that can be obtained from the scale is 46 and the maximum score is 230.
Wijma Birth Expectation/ Experience Scale-A Version | 12 weeks
  0 is expressed as "completely" and 5 is expressed as "none". While the minimum score on the scale is 0, the maximum score is 165.

SECONDARY OUTCOMES:
Psychosocial Health Assessment Scale in Pregnancy sub-dimensions | 12 weeks
  In the scale, the first sub-dimension evaluates "Characteristics of pregnancy and spousal relationship", the second sub-dimension evaluates "Characteristics of anxiety and stress", the third sub-dimension evaluates "Characteristics of domestic violence", the fourth sub-dimension evaluates "Characteristics of psychosocial support need", the fifth sub-dimension evaluates "Family characteristics" and the items in the sixth sub-dimension evaluates "Characteristics of physical-psychosocial changes related to pregnancy". scale, it is stated that each item should be scored between 1-5 (1= Not at all, 2= A little, 3= Moderately, 4= A lot, 5= Very much). The minimum score that can be obtained from the scale is 46 and the maximum score is 230.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Univeristy, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THERE IS ONE AUTHOR.